CLINICAL TRIAL: NCT05751356
Title: A Phase I Study to Evaluate the Safety, Tolerability and Pharmacokinetics of TR128 in Patients With Advanced Solid Tumors
Brief Title: TR128 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Tarapeutics Science Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TR128-CN-PI-01
Record Dates: First submitted 2023-02-20; First posted 2023-03-02 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Intervention Model Description: Dose escalation and expansion
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TR128 (Experimental)
  Interventions: Drug: TR128

INTERVENTIONS:
Drug: TR128 — TR128 will be given daily for 28 days in 28-day cycles until there appears evidence of progressive disease, intolerable toxicity, or the subject discontinues from the study treatment for other reasons. Starting dose is 100mg, with escalation to 500mg.

SUMMARY:
This is a open-label, 3+3 design, dose escalation and expansion, phase I study, to evaluate the safety and tolerability, and to determine the Recommended Phase II Dose (RP2D) of TR128 when administered qd in patients with advanced solid tumors. Up to 5 cohorts of 3-6 patients each will be treated in dose escalation phase of the study. One cycle is 28 days. Dose expansion phase to further evaluate the safety, tolerability and preliminary anti-tumor activity of TR128 at the RP2D.

DETAILED DESCRIPTION:
This phase I study of TR128 will investigate the tolerability, safety, pharmacokinetics (PK) and preliminary efficacy of TR128, and will define the maximum tolerated dose (MTD) of TR128 using 3+3 design. A dose expansion phase will identify the recommended phase 2 dose. In this clinical study, TR128 is given orally daily. A treatment cycle is defined as 28 days. Patients will receive study treatment until criteria for study termination are met. A safety follow-up visit will be conducted 28 days after the last dose of study treatment. Patients who discontinue study treatment for reasons other disease progression will have post-treatment follow-up for disease assessment until start of new anticancer treatment, patient withdraws consent, is lost to follow-up, death, or until the sponsor stops the study, whichever comes first.

Adverse events (AEs) will be assessed using the NCI Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0.

Tumor response will be assessed by computed tomography (CT) and /or magnetic resonance imaging (MRI) scan using RECIST1.1 criteria, assessed by the investigator.

ELIGIBILITY:
Inclusion Criteria:

* fully understand the procedures of the clinical study and participate voluntarily with signed and dated written informed consent form, comply with the requirements of the study protocol.
* males and/or females at least 18 years old when signing the informed consent form.
* histologically or cytologically confirmed patients with advanced malignant solid tumors, eligible patients must have failed standard treatment, no standard treatment, or not suitable for standard treatment at this stage as determined by the investigator.
* measurable disease with at least one lesion amenable to response assessment per RECIST 1.1.
* eastern cooperative oncology group performance status (ECOG) ≤1 at screening.
* life expectancy of at least 3 months.
* acceptable organ function: Absolute neutrophil count(ANC)≥1.5×109/L; Platelet count(PLT)≥90×109/L; Hemoglobin(Hb)≥90 g/L; International Normalized Ratio (INR) or Prothrombin Time (PT)≤1.5×Upper limit of normal value (ULN), Activated Partial Thromboplastin Time (APTT)≤1.5×ULN ; Total bilirubin(TBIL)≤1.5×Upper limit of normal value(ULN) (≤3× ULN if there is liver involvement); Alanine aminotransferase(ALT)≤2.5×ULN and aspartate aminotransferase(AST)≤2.5×ULN (≤ 5 × ULN if there is liver involvement); Creatinine (Cr) ≤1.5×ULN or Creatinine Clearance (CCr) ≥50 ml/min (calculated by Cockcroft-Gault formula).
* fertile male and female must agree to use medically approved contraceptives during the study and within 6 months after the last dose of the study.

Exclusion Criteria:

* medical history and surgical history excluded according to the protocol.
* any previous medical treatment history exclude from the protocol.
* abnormal laboratory results exclude from the protocol.
* pregnant and lactating women (currently breast-feeding or less than six months after delivery although not breast-feeding).
* unsuitable for the study by the investigator's judgment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Adverse Events and Serious Adverse Events | from the first dose to within 30 days after the last dose
  Frequency, duration, and severity of Adverse Events and Serious Adverse Events evaluated by NCI CTCAE v5.0
Dose limited toxicities | within 28 days after the first dose
  Incidence of dose limited toxicities
Maximum tolerated dose | Throughout the study for approximately 2 years
  Evaluated by safety review committee
Recommended phase II dose | Throughout the study for approximately 2 years
  Evaluated by safety review committee

SECONDARY OUTCOMES:
AUClast | within 31 days after the first dose
  Characterize the pharmacokinetic profile of TR128
AUCinf | within 31 days after the first dose
  Characterize the pharmacokinetic profile of TR128
Cmax | within 31 days after the first dose
  Characterize the pharmacokinetic profile of TR128
Tmax | within 31 days after the first dose
  Characterize the pharmacokinetic profile of TR128
CL/F | within 31 days after the first dose
  Characterize the pharmacokinetic profile of TR128
Vz/F | within 31 days after the first dose
  characterize the pharmacokinetic profile of TR128
Terminal half-life (T1/2) | within 31 days after the first dose
  Characterize the pharmacokinetic profile of TR128
ORR | throughout the study for approximately 2 years
  Efficacy-overall response rate
PFS | throughout the study for approximately 2 years
  Efficacy-progression free survival
DOR | throughout the study for approximately 2 years
  Efficacy-duration of response
DCR | throughout the study for approximately 2 years
  Efficacy-disease control rate

CONTACTS AND LOCATIONS:
Overall Officials: Lin Shen, MD, PhD, Principal Investigator — Peking University Cancer Hospital & Institute
Locations (3):
- China (3):
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - Harbin Medical University Cancer Hospital, Harbin, Heilonjiang
  - Tianjin Medical University Cancer Institute&Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No